CLINICAL TRIAL: NCT05672433
Title: Does the Bioactive Substance in Coffee, Cafestol, Have Preventive Properties on Type-2-diabetes? (Long-term Substudy)
Brief Title: Long-term Metabolic Effects of Cafestol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: cafestol.longterm
Record Dates: First submitted 2022-12-02; First posted 2023-01-05 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2022-06

CONDITIONS: Obesity, Abdominal
MeSH Terms: conditions — Obesity, Abdominal | interventions — cafestol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cafestol (Active Comparator): Participants in this arm ingest 6 mg cafestol capsules twice daily with breakfast and dinner.
  Interventions: Dietary Supplement: Cafestol
- Placebo (Placebo Comparator): Participants in this arm ingest placebo capsules twice daily with breakfast and dinner.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Placebo — Capsule without cafestol twice daily
  Arms: Placebo
Dietary Supplement: Cafestol — Capsule with 6 mg cafestol twice daily
  Arms: Cafestol

SUMMARY:
Twelve-week double-blinded, placebo-controlled, parallel intervention study on 40 participants with a large waist circumference who will ingest cafestol or placebo capsules twice daily. Insulin resistance is measured before and after the twelve-week intervention.

DETAILED DESCRIPTION:
Participants are randomly allocated to the cafestol intervention group or placebo group. Before and after the twelve-week intervention the participants partake in:

* A modified two-stage Insulin Suppression Test to determine insulin mediated glucose uptake. Fasting participants receive body-surface-area-adjusted octreotide, insulin and glucose infusions for 240 minutes. Octreotide is infused with the same rate throughout the test. Insulin and glucose infusions are slow for the initial 120-minute stage and increased the final 120-minute stage, simulating fasting and post-postprandial conditions, respectively. Steady state measurements of plasma glucose are acquired the final 30 minutes of each stage, at time points 100, 110, 120, 220, 230 and 240 minutes.
* A mixed meal test. Fasting participants consume 75 g. white bread, 10 g. butter, 30 g. cheese and 200 ml. orange juice. Blood samples are drawn at time points -15, 0, 15, 30, 60, 90, 120, 180 and 240 min for glucose-, insulin-, glucagon- and triglyceride measurements.
* A Magnetic Resonance Imaging (MRI) scan. Participants undergo dixon-sequences scanning the abdomen, assessing visceral and sub-cutaneous fat volume and liver fat content. Magnetic Resonance (MR) spectroscopy is also used to determine fat percentage of the liver.
* 24-hour ambulatory blood pressure measurement, every 20 minutes during daytime and every 30 minutes during nighttime.
* 1-week continuous glucose measurement using blinded continuous glucose monitor/sensor on upper arm.
* Fecal and urine sampling
* 72-hour food-diary
* Fasting blood samples:

  * Insulin, c-peptide, HbA1c and glucose
  * Total cholesterol, high density lipoprotein (HDL), low density lipoprotein (LDL) and triglycerides
  * Thyroid-stimulating hormone (TSH)
  * Alanine aminotransferase, creatinine, sodium and potassium
  * High sensitivity C reactive protein (CRP) and alpha-hydroxybutyrate
  * C-terminal telopeptide (CTX) and Procollagen type 1 N-terminal propeptide (P1NP)
  * Parathyroid hormone (PTH), Vitamin D and Ionized calcium
  * Monocyte Chemoattractant Protein-1 (MCP-1)
  * Interleukin 1 & 8 (IL-1α, IL-1β, IL-8)
  * Gastric inhibitory polypeptide (GIP), Glucagon-like peptide-1 (GLP-1) and Glucagon- like peptide-2 (GLP-2)
  * Growth/differentiation factor 15 (GDF-15)
  * Tumor necrosis factor (TNFα)
  * Fasting assessment of insulin resistance (Homeostatic Model Assessment for Insulin Resistance by C-peptide).

Pre-intervention and end-intervention test results will be compared using repeated-measures ANOVA / mixed models.

ELIGIBILITY:
Inclusion Criteria:

Waist circumference > 102 cm (men) / 88 cm (women)

Exclusion Criteria:

* Type 2 diabetes (HbA1c > 48 mmol/mol) or in treatment with antidiabetic drugs
* Pregnancy
* Planned pregnancy
* Breastfeeding
* Significant comorbidity expected to unable the subject from completing visits

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06-28 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Steady state plasma glucose during stage 2 of insulin suppression test (mmol/L) | 220, 230 and 240 minutes after test-start. Comparison between pre-intervention and end-intervention steady state plasma glucose.
  Subjects are administered a 25 μg octreotide bolus at time-point 0 minutes and subsequently infused with 0.27 μg octreotide / m2 • minute, 6 milliunits (mU) insulin / m2 • minute, and 50 mg glucose / m2 • minute. At time-point 120 minutes, infusion speeds were increased to to 32 mU insulin / m2 • minute and 267 mg glucose / m2 • minute.
Steady state plasma glucose during stage 1 of insulin suppression test (mmol/L) | 100, 110 and 120 minutes after test-start. Comparison between pre-intervention and end-intervention steady state plasma glucose.
  Subjects are administered a 25 μg octreotide bolus at time-point 0 minutes and subsequently infused with 0.27 μg octreotide / m2 • minute, 6 mU insulin / m2 • minute, and 50 mg glucose / m2 • min.
Area under the curve for glucose during mixed meal test (mmol/L*min) | -15 to 240 minutes from ingestion of standardized meal at time point 0 minutes. Comparison between pre-intervention and end-intervention area under the curves.
  Area under the curve for glucose during a mixed meal test.

SECONDARY OUTCOMES:
Area under the curve for insulin during mixed meal test (pmol/L*min) | -15 to 240 minutes from ingestion of standardized meal at time point 0 minutes. Comparison between pre-intervention and end-intervention area under the curves.
  Area under the curve for insulin during a mixed meal test.
Area under the curve for glucagon during mixed meal test (pmol/L*min) | -15 to 240 minutes from ingestion of standardized meal at time point 0 minutes. Comparison between pre-intervention and end-intervention area under the curves.
  Area under the curve for glucagon during a mixed meal test.
Area under the curve for triglycerides during mixed meal test (mmol/L*min) | -15 to 240 minutes from ingestion of standardized meal at time point 0 minutes. Comparison between pre-intervention and end-intervention area under the curves.
  Area under the curve for triglycerides during a mixed meal test.
Glycated hemoglobin (HbA1c) (mmol/mol) | 12-week change. Comparison between pre-intervention and end-intervention glycated hemoglobin levels.
  Glycated hemoglobin (HbA1c) (mmol/mol)
Liver fat content (%) | 12-week change. Comparison between pre-intervention scan and end-intervention scan.
  Measured with dixon-sequences scanning the abdomen and MR-Spectroscopy.
Visceral fat content (ml) | 12-week change. Comparison between pre-intervention scan and end-intervention scan.
  Measured with dixon-sequences scanning the abdomen
Subcutaneous fat content (ml) | 12-week change. Comparison between pre-intervention scan and end-intervention scan.
  Measured with dixon-sequences scanning the abdomen
One-week continuous glucose measurement | Average glucose measured every 15 minutes for one week prior to study day 1 and 3. 12-week change. Comparison between pre-intervention measurement and end-intervention measurement.
  One-week continuous glucose measurement data.
Blood pressure (mmHg) | 12-week change. Comparison between pre-intervention average ambulatory blood pressure and end-intervention average ambulatory blood pressure.
  Average daytime and night-time ambulatory blood pressure. 24-hour ambulatory blood pressure measurement, measured every 20 minutes during daytime and every 30 minutes during nighttime.
Food consumption in kilocalories (kcal) | 12-week change. Comparison between pre-intervention food consumption and end-intervention food consumption.
  Food consumption is registered for 72-hours prior to study day 1 and 3. Food consumption is measured in kilocalories (kcal).

OTHER OUTCOMES:
Fasting glucose (mmol/l) | Measured on study day 1 and 3. 12-week change. Comparison between pre-intervention blood samples and end-intervention blood samples.
Fasting insulin (pmol/l) | Measured on study day 1 and 3. 12-week change. Comparison between pre-intervention blood samples and end-intervention blood samples.
Fasting total cholesterol (mmol/l), | Measured on study day 1 and 3. 12-week change. Comparison between pre-intervention blood samples and end-intervention blood samples.
Fasting HDL (mmol/l) | Measured on study day 1 and 3. 12-week change. Comparison between pre-intervention blood samples and end-intervention blood samples.
Fasting LDL (mmol/l) | Measured on study day 1 and 3. 12-week change. Comparison between pre-intervention blood samples and end-intervention blood samples.
Fasting triglycerides (mmol/l) | Measured on study day 1 and 3. 12-week change. Comparison between pre-intervention blood samples and end-intervention blood samples.
Fasting thyroid-stimulating hormone (international unit (IU)/l) | Measured on study day 1 and 3. 12-week change. Comparison between pre-intervention blood samples and end-intervention blood samples.
Fasting alanine aminotransferase (unit(U)/l) | Measured on study day 1 and 3. 12-week change. Comparison between pre-intervention blood samples and end-intervention blood samples.
Fasting high sensitivity c reactive protein (mg/l) | Measured on study day 1 and 3. 12-week change. Comparison between pre-intervention blood samples and end-intervention blood samples.
Fasting alpha-hydroxybutyrate (mmol/l) | Measured on study day 1 and 3. 12-week change. Comparison between pre-intervention blood samples and end-intervention blood samples.
Fasting C-terminal telopeptide (µg/l) | Measured on study day 1 and 3. 12-week change. Comparison between pre-intervention blood samples and end-intervention blood samples.
Fasting procollagen type 1 N-terminal propeptide (µg/l) | Measured on study day 1 and 3. 12-week change. Comparison between pre-intervention blood samples and end-intervention blood samples.
Fasting parathyroid hormone (pmol/l) | Measured on study day 1 and 3. 12-week change. Comparison between pre-intervention blood samples and end-intervention blood samples.
Fasting vitamin D (nmol/l) | Measured on study day 1 and 3. 12-week change. Comparison between pre-intervention blood samples and end-intervention blood samples.
Fasting ionized calcium (mmol/l) | Measured on study day 1 and 3. 12-week change. Comparison between pre-intervention blood samples and end-intervention blood samples.
Fasting monocyte chemoattractant protein-1 (pg/ml) | Measured on study day 1 and 3. 12-week change. Comparison between pre-intervention blood samples and end-intervention blood samples.
Fasting interleukin 1 (pg/ml) | Measured on study day 1 and 3. 12-week change. Comparison between pre-intervention blood samples and end-intervention blood samples.
Fasting interleukin 8 (pg/ml) | Measured on study day 1 and 3. 12-week change. Comparison between pre-intervention blood samples and end-intervention blood samples.
Fasting gastric inhibitory polypeptide (pmol/l) | Measured on study day 1 and 3. 12-week change. Comparison between pre-intervention blood samples and end-intervention blood samples.
Fasting glucagon-like peptide-2 (pmol/l) | Measured on study day 1 and 3. 12-week change. Comparison between pre-intervention blood samples and end-intervention blood samples.
Fasting growth/differentiation factor 15 (ng/l) | Measured on study day 1 and 3. 12-week change. Comparison between pre-intervention blood samples and end-intervention blood samples.
Fasting tumor necrosis factor (TNFα) | Measured on study day 1 and 3. 12-week change. Comparison between pre-intervention blood samples and end-intervention blood samples.
Fasting Homeostatic Model Assessment for Insulin Resistance by C-peptide (arbitrary unit). | Measured on study day 1 and 3. 12-week change. Comparison between pre-intervention blood samples and end-intervention blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Søren Gregersen, M.D. Ph.D, Principal Investigator — Aarhus University Hospital
Locations (1):
- Steno Diabetes Center Aarhus, Aarhus, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No